CLINICAL TRIAL: NCT03033862
Title: Thrombogenicity Assessment in Patients Treated With Bioresorbable Vascular Scaffolds
Status: Withdrawn | Type: Observational
Why Stopped: Stent taken off market due to safety concerns
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2565
Record Dates: First submitted 2017-01-06; First posted 2017-01-27 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intervention with Bioresorbable Vascular Scaffold: Implant of Abbott Bioresorbable stent
  Interventions: Device: Bioresorbable Vascular Scaffold
- Intervention with Drug Eluting Stent: implant of drug eluting stent
  Interventions: Device: Drug Eluting Stent

INTERVENTIONS:
Device: Bioresorbable Vascular Scaffold — Bioresorbable Vascular Scaffold
  Groups: Intervention with Bioresorbable Vascular Scaffold
Device: Drug Eluting Stent — Drug Eluting Stent
  Groups: Intervention with Drug Eluting Stent

SUMMARY:
Platelet activation and aggregation, intrinsic thrombogenicity, and biomarkers (fibrinogen, C-reactive protein, platelet endothelial cell adhesion molecule, von Willebrand factor, p-selectin) will be measured and compared following the implantation of Bioreabsorbable Vascular Scaffolds and Drug Eluting Stents.

ELIGIBILITY:
Inclusion Criteria:

1. Subject may be of either sex and of any race, and must be >18 years of age.
2. Subjects undergoing elective PCI due to de novo native coronary artery lesions (length ≤24 mm) with a reference vessel diameter of ≥2.5 mm and ≤3.75 mm.
3. Subject agrees to not participate in any other investigational or invasive clinical study for a period of 3 months following the index procedure.
4. Subject must be willing and able to give appropriate informed consent.
5. The subject is able to read and has signed and dated the informed consent document including authorization permitting release of personal health information approved by the investigator's Institutional Review Board (IRB).

Exclusion Criteria:

* Hemodynamically unstable at the time of enrollment.
* Concurrent or anticipated treatment with warfarin (or derivatives, e.g., phenprocoumon), oral factor Xa inhibitor, or oral direct thrombin inhibitor after enrollment.
* GPI use prior to or at the time of PCI.
* History of a bleeding, or evidence of active abnormal bleeding.
* History at any time of intracranial hemorrhage, intracranial or spinal cord surgery, or a central nervous system tumor or aneurysm.
* Documented sustained severe hypertension (systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg) at enrollment.
* Severe valvular heart disease, as defined by the American College of Cardiology /American Heart Association.
* History within 30 days before enrollment of invasive surgeries (other than mentioned above), or is anticipating one during the course of their study participation, or is planning to have one within 1 month post dosing with the study drug.
* History within 30 days before enrollment of TIA and ischemic (presumed thrombotic) stroke/CVA.
* Known platelet count <100,000/mm3 within 30 days before enrollment.
* Known active hepatobiliary disease, or known unexplained persistent increase in serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) activity to two times or more the upper limit of the reference range (upper limit of "normal" [↑2xULN]).
* Any serious medical comorbidity (e.g., active malignancy) such that the subject's life expectancy is <24 months.
* Known current substance abuse at the time of enrollment.
* Current participation in any other study of investigational therapy or participation in such a study within the last 30 days.
* Known hypersensitivity to any component of the current investigational product.
* Female subject of child-bearing potential.
* Subject is a woman who is breast-feeding.
* Subject is part of the staff personnel directly involved with this study or is a family member of the investigational staff.
* LVEF <30%
* Subject with known renal insufficiency with an estimated GFR <30 ml/min/1.73m or dialysis at the time of screening
* Subject requiring at least two lesion treatment and more suitable for staged PCI.
* Moderate or heavy calcification, tortuosity or other conditions are present proximal or within the target segment, reducing the likelihood that the Absorb BVS or XIENCE can be either delivered to or expanded at the lesion.
* Extreme angulation (≥90°) proximal to or within the target lesion.
* Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
* Lesion located within or distal to a diseased arterial graft or SVG.
* Aorto-ostial lesion (within 3 mm of the aorta junction).
* Lesion located in the left main artery.
* Lesion located within 2 mm of the origin of the LAD or LCX.
* Lesion involving a bifurcation with a:

  * side branch ≥ 2 mm in diameter, or
  * side branch with either an ostial or non-ostial lesion with diameter stenosis > 50%, or
  * side branch requiring dilatation.
* Target vessel contains thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include subjects with stable ischemic heart disease receiving percutaneous coronary intervention.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Thrombogenicity from baseline after device implantation | 60 Days
  Platelet activation and aggregation, intrinsic thrombogenicity, and biomarkers will be measured at baseline and then reassessed at multiple time points after the implantation of the study device.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Gurbel, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States